CLINICAL TRIAL: NCT05244031
Title: Intraoperative Placement of Superficial Erector Spinae Plane Block in Spine Surgery; An Effective Approach at Enhanced Recovery After Spine Surgery
Brief Title: Intraoperative Placement of Superficial Erector Spinae Plane Block; A New Approach in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-271
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Pain; Spine Deformity; Spine Injury; Spine Fracture; Spine Malformation
Keywords: Postoperative pain; Superficial Erector Spinae Plane Block; Spine Surgery; Local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Spinal Injuries; Spinal Fractures | interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial ESP (Active Comparator): The investigators performed superficial erector spina plane block to that patient group for postoperative analgesia
  Interventions: Procedure: superficial erector spina plane block
- Control group (Active Comparator): The investigators performed intravenous opioid infusion with PCA to that patient group for postoperative analgesia
  Interventions: Procedure: Standard (opioid-based) analgesia

INTERVENTIONS:
Procedure: superficial erector spina plane block — The investigators performed superficial erector spina plane block to that patient group for postoperative analgesia
  Arms: Superficial ESP
Procedure: Standard (opioid-based) analgesia — The investigators performed intravenous opioid infusion with PCA to that patient group for postoperative analgesia
  Arms: Control group

SUMMARY:
Major spine surgery causes severe postoperative pain. The primary objective of this randomized controlled study is to compare the effect of ultrasound (US)-guided superficial erector spinae plane (ESP) block on 48-hour postoperative cumulative opioid requirements with standard (opioid-based) analgesia.

DETAILED DESCRIPTION:
46 patients (ASA I-II-III) between 18 and 65 years of age, who were to undergo spine surgery, were randomized and divided into two groups. (23 patients in each of the control and superficial ESP groups). Superficial ESP block was performed for SESP group and standard (opioid-based) analgesia performed in the control group. Postoperative analgesia was provided by intravenous morphine infusion using a patient-controlled analgesia device. Postoperative numeric rating scale values were the primary outcome measure. 24-hour total morphine consumption was secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65
* Patients who will undergo spine surgery (at least two level)
* ASA I-II-III patients

Exclusion Criteria:

* Clinically known local anesthetic allergy
* Morbid obesity (body mass index>40 kg m2)
* Clinically diagnosis of opioid, alcohol and substance dependence
* Clinically diagnosis of psychiatric disease
* Coagulopathy
* Patients with ASA IV-V
* Single level surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
NRS scores of patients | 48 hours postoperatively
  NRS at 1, 6,12, 18, 24, 36, 48th hours

SECONDARY OUTCOMES:
Postoperative 48-hours total morphine consumption | 48 hours postoperatively
  This will be measured only one time by pca device at the 48th hour after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)